CLINICAL TRIAL: NCT05903651
Title: Retinal Deep PhenotypingTM by a Novel Mydriatic Hyperspectral Retinal Camera (MHRC) and Analysis by Deep Learning
Brief Title: Retinal Deep PhenotypingTM
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-002
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Group Assignment: The subjects will undergo a single retinal imaging session with the Optina MHRC device, on one or both eyes.

SUMMARY:
This study aims to collect a baseline dataset of MHRC retinal scans that will be used for the pre-training of deep learning models from the hyperspectral retinal image phenotypic features that may form the basis for multiple future classification applications. A sub-set of the images will also be analyzed by eye specialists to determine if visual inspection of the images could provide useful information in their practice.

As an exploratory study, there are no endpoints per se, however the following sub-objective will be evaluated for determining the success of this study:

* Collection and characterization of MHRC retinal images from at least 2000 participants that score at least 80 on the real-time Quality Index (included in the MHRC software).
* Development of at least one (1) DL model of the retina. Models may be used for the development of novel classifier tests and potential use in a clinical setting.
* At least 5% of participants shall have an MHRC retinal image reviewed by an eye specialist (Optometrist or Ophthalmologist) to assess the image quality and potential clinical usefulness.

DETAILED DESCRIPTION:
This is an exploratory, observational, cross-sectional, multi-site study designed to collect a baseline dataset of MHRC retinal image scans for use in Deep Learning models and to determine the feasibility of visual inspection of the images for use in Optometry and/or Ophthalmology clinical practice. Subjects will be recruited from eye clinics where patients will undergo mydriasis (pupil dilation) as part of their clinical visit. Eligible participants will be provided information about the study and delegated site personnel will assist with the Informed Consent process. If a participant provides their Informed Consent, they will be enrolled in the study and undergo a single retinal imaging session with the Optina MHRC device, on one or both eyes.

The MHRC retinal images will be transferred to a Picture Archiving and Communication System (PACS) for archiving and later evaluation. Additional information about the Study Participant will be captured in an Electronic Data Capture (EDC) system, including age, date of birth, gender, race/ethnicity, and color of their iris.

Images will be transferred to Optina for further digital analysis, including pre-processing (normalization, registration, and segmentation), feature extraction, and inclusion in Deep Learning models.

A subset (at least 5%) of the MHRC retinal scans will undergo visual inspection by an eye specialist (Ophthalmologist or Optometrist) to determine their quality and utility for inclusion in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

• Adults 18 years and older who will undergo mydriasis (pupil dilation) as part of their eye clinic visit.

Exclusion Criteria:

* Pupil dilation contraindicated (due to a pathology, or presence of 3 quadrants with Van Herick grading of 0 or 1 without iridotomy).
* Inadequate pupil dilatation (< 6mm diameter) preventing uniform illumination of the retina with the MHRC.
* Refractive error outside the range of -15 D to +15 D.
* Deficient visual fixation (inability to fixate for at least 2 s)
* Inability of obtaining at least 3 images of satisfactory quality with the MHRC per the Optina Diagnostics quality index software and /or per the eye specialists' evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 years and older who have undergone pupil dilation and are not contraindicated for mydriatic imaging with a fundus camera. Ideally, the study population will be reflective of the adult population with the following estimates for demographics.
  Gender* 49% Male 51% Female
  Age* 45% 18-44 years old 55% 44+ years old
  Ocular Health ǂ 70% Normal ocular health 30% Eye symptoms
  * based on 2021 Canada census data ǂ based on CNIB Fast Facts about Vision Loss
Sampling Method: Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
At least one (1) pre-trained DL model from hyperspectral retinal images. | 12 months
Report describing the clinical utility of visual inspection of the MHRC retinal images. | 12 months
Review of any safety events (AE, SAE, UADEs) that occur throughout the study. | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Ecole d'Optometrie, University of Montreal, Montreal, Quebec
  - Clinique d'Opthalmologie desLaurentides, Institue de l'Oeil (IOL), Montreal, Quebec